CLINICAL TRIAL: NCT03355833
Title: Comparing Prognostic Performance of SEPSIS 2 and SEPSIS 3 Strategies at the Emergency Service
Acronym: StraSEP
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Responsible Party: Sponsor
Other Study IDs: 2016-05Obs-CHRMT
Record Dates: First submitted 2017-11-20; First posted 2017-11-28 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2017-11

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In 2016, the Third International Consensus proposed a new strategy to screen aggravating risk in patients with septic shock. This strategy is based on quick-SOFA and the SOFA score. The main objective is to compare the prognostic performance of SEPSIS 3 against the previous strategy SEPSIS 2 to predict the admission in intensive care unit or the intra-hospital death.

DETAILED DESCRIPTION:
This study compare the prognostic performance of two strategies. It's a monocentric, retrospective study in patients admitted to the emergency department.

ELIGIBILITY:
Inclusion Criteria:

* Aged of 18 years or more
* Initiation of one or more antibiotics in the Accident and Emergency Department in the Metz-Thionville hospital (CHR) site Mercy, for curative purpose, regardless of the infectious aetiology
* Hospitalized in the CHR Metz-Thionville thereafter

Exclusion Criteria:

* Minors patients
* Absence of antibiotic treatment initiated in the Emergency department
* Prescription of antibiotic treatment in the emergency department for preventive purpose
* Transferred by hospitalisation service of CHR Metz-Thionville in the emergency department
* Absence of hospitalisation following their passage through the emergency department
* Transferred to hospitalisation in an other establishment
* Presence, at the admission, of an antibiotic treatment
* Patients deceased in the emergency department

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Retrospective study in patients admitted to the emergency department in the CHR Metz-Thionville
Sampling Method: Probability Sample
Enrollment: 228 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Intrinsic and Extrinsic properties of SEPSIS 3 strategy | Day 1
  The percentage of patients with high qSOFA score (2 or more) who were admitted in intensive care unit or who have died during their stay in hospital and rather the percentage of patients with a small qSOFA score who survived without passing through intensive care unit

SECONDARY OUTCOMES:
Correlation between lactate levels and mortality | Day 1
  lactate levels at their admission